CLINICAL TRIAL: NCT06281613
Title: Comparison of AMCOP Bioactivator and High-pull Headgear in Treating Skeletal Class II Hyperdivergent Pediatric Patients: a Retrospective Study
Brief Title: Comparison of AMCOP Bioactivator and High-pull Headgear in Treating Skeletal Class II Hyperdivergent Pediatric Patients
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Other Study IDs: 2024-AMCOPTEO
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Skeletal Malocclusion
Keywords: hyperdivergency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group
  Interventions: Device: AMCOP group
- Control Headgear
  Interventions: Device: High-pull headgear

INTERVENTIONS:
Device: AMCOP group — Patients were treated with AMCOP for 18 months.
  Groups: Case group
Device: High-pull headgear — Patients were treated with high-pull headgear for 18 months.
  Groups: Control Headgear

SUMMARY:
The aim of the present study was to retrospectively compare the clinical use of high-pull headgear versus AMCOP bioactivators for hyperdivergent pediatric patients.

Cephalometric radiographs from pediatric patients treated at the Unit of Orthodontics and Pediatric Dentistry, Section of Dentistry, Department of Clinical, Surgical, Diagnostic and Pediatric Sciences, University of Pavia, Pavia, Italy and at the private practice of Dr. Cardarelli, Isernia, Italy will be collected.

Cephalometric tracing from Giannì analysis will be performed at the baseline (T0) and after 18 months of treatment (T1).

DETAILED DESCRIPTION:
The aim of the present study was to retrospectively compare the clinical use of high-pull headgear versus AMCOP bioactivators for hyperdivergent pediatric patients.

Cephalometric radiographs from pediatric patients treated at the Unit of Orthodontics and Pediatric Dentistry, Section of Dentistry, Department of Clinical, Surgical, Diagnostic and Pediatric Sciences, University of Pavia, Pavia, Italy and at the private practice of Dr. Cardarelli, Isernia, Italy will be collected.

Cephalometric tracing from Giannì analysis will be performed at the baseline (T0) and after 18 months of treatment (T1).

ELIGIBILITY:
Inclusion Criteria:

* mixed or permanent dentition
* skeletal class II malocclusion diagnosed with ANB angle > 4° from cephalometric radiograph
* skeletal hyperdivergency calculated from AnsPns^GoGn angle > 25°, and at least S-Ar^Go > 149° or Ar-Go^Gn > 137°

Exclusion Criteria:

* lack of compliance in the use of the orthodontic appliance
* syndromic patients, cleft lip or cleft palate, severe malformations and asymmetries of the jaws.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Orthodontic patients
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change in cephalometric angular measurements | Baseline (T0) and after 18 months (T1)
  The following angular measurements will be calculated in cephalometric radiographs:
  SNA SNB ANB SN^GoGn AnsPns^GoGn Occl-MP Occl-AnsPns N-S-Ar S-Ar-Go Ar-Go-N N-Go-Gn 11-occl 11-ANSPNS 41-occl 41-GoGn Nasolabial angle Facial angle
Linear regressions | Baseline (T0) and after 18 months (T1)
  Linear regressions among the variables of the study and sex, age, and group of the patients will be performed.
Change in cephalometric linear measurements | Baseline (T0) and after 18 months (T1)
  The following linear measurements will be calculated in cephalometric radiographs:
  Anterior cranial base Mandibular body Mandibular ramus Posterior facial height Anterior facial height A0B0

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Mac, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.